CLINICAL TRIAL: NCT05386875
Title: Evaluation of rK28 RDT for the Diagnosis of Visceral Leishmaniasis in Kenya, Towards Strengthening Recommendations for Its Use and Access in Eastern Africa
Brief Title: Evaluation to Assess the Usability of rK28 for the Diagnosis of Visceral Leishmaniasis in Kenya
Acronym: rK28-AccDemo
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Foundation for Innovative New Diagnostics, Switzerland (Other)
Collaborators: Kenya Medical Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: NT012
Record Dates: First submitted 2022-04-21; First posted 2022-05-23 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Visceral Leishmaniasis
MeSH Terms: conditions — Leishmaniasis, Visceral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood collection is part of the routine sampling procedure for VL diagnosis. Blood will be collected into heparinized tubes and tested immediately or stored at 4⁰C until used. Serum will be separated once blood aliquots are prepared (this is optional for this study, contingent on availability of tests). Dry blood spot (DBS) will also be collected for DAT testing. Blood aliquots, serum and DBS samples will be stored at -20⁰C at the study facility and later transferred to KEMRI, up to a maximum of 5 years. Stored samples will serve for quality control (QC) purposes.
  The transfer of samples to any institution outside Kenya is not expected in this study. In the event that this may be required, the legal transfer will be regulated by material transfer agreements (MTA) or equivalent documents provided by FIND
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: rK28 — rK28 RDT (Index): The Leishmania Ab Rapid Test is a rapid immunochromatographic test that uses the recombinant antigen rK28 to detect antibodies against Leishmania species in human serum, plasma, or whole blood samples intended for primary VL diagnosis. It is a Research Use Only product commercialized by CTK Biotech, Inc. (USA).
  IT-Leish rK39 RDT: Rapid immunochromatographic test for detection of antibodies against Leishmania species in human serum, plasma, or whole blood samples of utility in the VL diagnosis algorithm. It is a CE marked product commercialized by Bio-Rad (France). This is currently the recommended RDT for VL diagnosis in Kenya.
  Kalazar Detect rK39, RDT: Rapid immunochromatographic test for detection of antibodies against Leishmania species in human serum, plasma, or whole blood samples of utility in the VL diagnosis algorithm. It is a CE marked product commercialized by InBios (United States).
  Other Names: IT-Leish rK39; KalazarDetect rK39

SUMMARY:
Visceral leishmaniasis (VL) is a fatal disease caused by Leishmania parasites and transmitted by female phlebotomine sandflies. The disease is a serious public health problem in eastern Africa; including Kenya where an estimated 4000 cases occur annually and 5 million people are at risk of infection. Accurate diagnosis of VL is critical for appropriate treatment. Currently, VL diagnosis in Kenya is based on testing suspected patients with the IT-Leish rK39 rapid diagnostic test (RDT) followed by other tests such as the Direct Agglutination Tests (DAT) and microscopy of tissue aspirates (splenic, bone marrow, lymph node) on rK39-negative patients. However, these diagnostic tools present several challenges including; the need for expertise, equipment and low diagnostic sensitivity of (85%) for DAT and rK39. Alternative VL diagnostic tools that are readily available, easy to use with increased sensitivity are needed to improve VL surveillance and control in Kenya. In the present study, we will assess rK28 as a diagnostic tool including performance with increased sensitivity when used together with IT-Leish rK39 and its potential for inclusion in VL diagnosis algorithms and evaluate Kala-azar Detect rK39 for potential use in Kenya. Suspected patients presenting at VL testing facilities in Marsabit, Turkana and Wajir Counties will be recruited prospectively and tested using IT-Leish rK39 followed by DAT for case confirmation according to the national guidelines. Alongside the case confirmation, samples from participants will also be tested using the rK28 and Kala-azar Detect rK39 in whole blood and serum. The collected data will be analyzed and compared separately between the RDTs as well as in combination, and the performance of the algorithms determined retrospectively. This design will enable the assessment of the sensitivity of combining rK28 and rK39 (Kala-azar Detect) compared to rK39 (IT-Leish/Kala-azar Detect) alone. Microscopy will be used as confirmatory test. We will also assess the feasibility, usefulness, and cost-effectiveness of rK28 in the VL diagnostic algorithm, through sensitivity analyses. The improved understanding of rK28 as a VL diagnostic tool and its potential for inclusion in the VL diagnosis algorithm could enable faster and more effective management of cases and accelerate elimination of VL.

ELIGIBILITY:
Inclusion Criteria:

* All patients ≥ 1 year, with clinical signs and symptoms compatible with VL (fever > 2 weeks, splenomegaly, wasting, malaria negative)
* Participants for whom written informed consent has been obtained (if aged 18 years and over) or signed by parents(s) or legal guardian for participants under 18 years of age. In the case of minors 12 - 17 years, assent from the children will to be obtained in addition to parental consent.

Exclusion Criteria:

* Relapse cases of VL (recrudescent infection 6-12 month after treatment).
* Participants with post-kala-azar dermal leishmaniasis
* Participants from whom, for any reason, the blood sample needed for the evaluation cannot be taken

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals presenting at health facilities in the participating sites or referred from peripheral health centres with suspicion of VL.
Sampling Method: Non-Probability Sample
Enrollment: 625 (Estimated)
Dates: Start 2022-12-31 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance | 12 months
  Sensitivity, Specificity, the negative and positive predictive values (NPV, PPV) along with their confidence intervals.
Diagnostic performance | 12 months
  Diagnostic odd ratio (DOR) or balanced Accuracy (BA).
Use cases | 12 months
  Use cases for the different combination of tests.

SECONDARY OUTCOMES:
Cost effectiveness | 12 months
  Cost estimates per test/algorithm
Access to diagnosis (optimum placement of RDTs) | 12 months
  Distance to the primary healthcare facility and to the referral facility.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Ndung'u, Principal Investigator — Find
Locations (4):
- Kenya (4):
  - Turkana County, Lodwar
  - Marsabit County, Marsabit
  - Kenya Medical Research Institute, Nairobi
  - Wajir County, Wajir